CLINICAL TRIAL: NCT00864032
Title: Phase I/II Trial of Neoadjuvant Conformal Radiotherapy Plus Sorafenib for Patients With Soft Tissue Sarcoma of the Extremity and Body Wall
Brief Title: Trial of Neoadjuvant Conformal Radiotherapy Plus Sorafenib for Patients With Soft Tissue Sarcoma of the Extremity and Body Wall
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Robert J. Canter, MD, Principal Investigator, University of California, Davis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STS Sorafenib; NCT00805727 (obsolete NCT alias)
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Results first posted 2013-04-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma of the extremity and body wall
MeSH Terms: conditions — Sarcoma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I (Experimental)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400mg twice daily
  Other Names: Nexavar

SUMMARY:
Patients will receive neoadjuvant sorafenib (investigational agent) in combination with preoperative external beam conformal radiotherapy (50 Gy in 25 fractions) for localized, large soft tissue sarcomas of the extremity and body wall prior to resection with curative intent. Sorafenib is an FDA-approved targeted agent for patients with renal cell carcinoma and hepatocellular carcinoma. Preliminary data suggest activity for sorafenib against soft tissue sarcoma in the metastatic setting. Limited data are available regarding the safety and efficacy of sorafenib in combination with radiotherapy.

The Phase I portion of the trial will seek to establish the safety of sorafenib and radiotherapy in the neoadjuvant setting for soft tissue sarcomas of the extremity and body wall. The Phase II portion of the trial will aim to determine the pathologic near-complete/complete response rate (≥ 95% tumor necrosis) of this multimodality therapy. Molecular and dynamic contrast-enhanced MRI studies will seek to establish correlative biological and imaging markers of response and/or resistance to this therapy.

DETAILED DESCRIPTION:
Patients will receive neoadjuvant sorafenib (investigational agent) in combination with preoperative external beam conformal radiotherapy (50 Gy in 25 fractions) for localized, large soft tissue sarcomas of the extremity and body wall prior to resection with curative intent. Sorafenib is an FDA-approved targeted agent for patients with renal cell carcinoma and hepatocellular carcinoma. Preliminary data suggest activity for sorafenib against soft tissue sarcoma in the metastatic setting. Limited data are available regarding the safety and efficacy of sorafenib in combination with radiotherapy.

The Phase I portion of the trial will seek to establish the safety of sorafenib and radiotherapy in the neoadjuvant setting for soft tissue sarcomas of the extremity and body wall. The Phase II portion of the trial will aim to determine the pathologic near-complete/complete response rate (≥ 95% tumor necrosis) of this multimodality therapy. Molecular and dynamic contrast-enhanced MRI studies will seek to establish correlative biological and imaging markers of response and/or resistance to this therapy.

Significant challenges exist in the treatment of patients with soft tissue sarcoma (STS) of the extremity and body wall. Major therapeutic goals for all patients include local disease-control, maximization of limb function, and avoidance of therapeutic morbidity. The standard approach for patients with STS has been based on radical resection with wide margins in combination with external beam radiation. Although local control rates in this setting range from 85 to 90%, patients remain at risk for substantial morbidity from this multimodality therapy. Furthermore, despite effective local therapy with surgery and radiation, approximately 50% of patients with high grade STS will die of disease within 5 years of diagnosis.

Experimental data and experience from other solid tumors suggest a significant synergistic effect when anti-angiogenic targeted therapies, such as sorafenib, are combined with radiotherapy (RT). Overproduction of angiogenic factors in the tumor vasculature leads to disordered/poorly regulated tumor perfusion which appears to normalize following delivery of anti-angiogenic agents. This, in turn, allows improved delivery of and susceptibility to cytotoxic agents, which is particularly important with RT since hypoxia is a key mechanism of resistance to this modality. Preliminary clinical data in rectal cancer and malignant brain tumors have demonstrated promising results from the combination of anti-angiogenic agents and RT with respect to downstaging of the primary tumor, local tumor control, and improved progression-free survival. Angiogenic factors are upregulated in patients with STS, and anti-angiogenic agents demonstrate activity against STS in the metastatic setting.

Consequently, we propose to evaluate preoperative combined modality sorafenib and conformal RT in patients with STS of the extremity and body wall in a prospective Phase I/II clinical trial. Key endpoints will be safety and toxicity in the Phase I trial and pathological response in the Phase II trial. Additional endpoints will include molecular and functional imaging correlative studies of biomarkers of response and resistance to treatment.

We hypothesize that this combination will be safe and will increase pathologic necrosis within the primary tumor at the time of surgical resection, translating into reduced volume of resected tissue, improved local disease-control, and ultimately improved disease-free survival. Functional imaging studies (dynamic contrast-enhanced MRI) and molecular examination of pre- and post-treatment tumor tissue and serum will allow correlation of changes in tumor blood flow, hypoxia transcription factors, phosphorylated ERK, and angiogenic markers to the degree of tumor necrosis following treatment with preoperative sorafenib and radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed soft-tissue sarcoma located on the extremity or body wall.

  * Intermediate or High grade (NCI grade 2 or 3/3-tier system), > 5 cm in maximal dimension.
  * Low grade (NCI grade 1/3-tier system), > 8 cm in maximal dimension.
  * No evidence of regional or distant metastatic disease.
  * Patient must be 18 years of age or older.
  * Patient must have an ECOG performance status of ≤ 2.
  * Patient must have a histologic diagnosis of soft tissue sarcoma.
* Patient must have adequate bone marrow, liver, and renal function as assessed by the following:

  * Hemoglobin ≥ 9.0 g/dl
  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3.
  * Total bilirubin ≤ 1.5 mg/dL. NOTE: Patients with elevated bilirubin secondary to Gilbert's syndrome are eligible to participate in the study.
  * AST and ALT ≤ 2.5 times the institution upper limit of normal (ULN).
  * Creatinine ≤ 1.5 times ULN.
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the start of treatment . NOTE: Postmenopausal women must be amenorrheic for at least 12 months to be deemed not of reproductive potential.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.

Exclusion Criteria:

* Patient is receiving additional cancer-directed therapy at time of entry into trial.
* Patient has received or is receiving preoperative investigational treatment.
* Patient has congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Patient has history of cardiac ventricular arrhythmia requiring ongoing anti-arrhythmic therapy.
* Patient has uncontrolled hypertension, defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Patient has known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Patient has active clinically serious infection > CTCAE Grade 2.
* Patient has thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Patient has history of pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Patient has history of any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Patient has history of clinical or laboratory evidence of bleeding diathesis or coagulopathy.
* Patient has history of major surgery or significant traumatic injury within 4 weeks of first study drug.
* Patient has concomitant use of St. John's Wort or rifampin (rifampicin).
* Patient has known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Patient has any condition that impairs his or her ability to swallow whole pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Canter, MD, Principal Investigator — U C Davis Medical Center
Locations (1):
- University of california, Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Canter RJ, Borys D, Olusanya A, Li CS, Lee LY, Boutin RD, Christensen SD, Tamurian RM, Monjazeb AM. Phase I trial of neoadjuvant conformal radiotherapy plus sorafenib for patients with locally advanced soft tissue sarcoma of the extremity. Ann Surg Oncol. 2014 May;21(5):1616-23. doi: 10.1245/s10434-014-3543-7. Epub 2014 Feb 20. PMID 24554062

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib 200/200: Dose level 1 sorafenib 200 bid with concurrent neoadjuvant radiation therapy.
  sorafenib administered orally. agent administered during concurrent neoadjuvant radiation therapy. both modalities discontinued approximately 4 - 6 weeks prior to surgical resection with curative intent.
- Sorafenib 200/400: Dose level 2 sorafenib 200 mg PO Q AM and 400 mg PO Q PM with concurrent neoadjuvant radiation therapy.
  sorafenib administered orally. agent administered during concurrent neoadjuvant radiation therapy. both modalities discontinued approximately 4 - 6 weeks prior to surgical resection with curative intent.
  Traditional 3+3 dose escalation Phase I trial. Cohort 2 enrolled after completion of all 3 participants in dose level 1.
- Sorafenib 400/400: Dose level 3 sorafenib 400 mg PO BID with concurrent neoadjuvant radiation therapy.
  sorafenib administered orally. agent administered during concurrent neoadjuvant radiation therapy. both modalities discontinued approximately 4 - 6 weeks prior to surgical resection with curative intent.
Period: Overall Study
Arm/Group | Sorafenib 200/200 | Sorafenib 200/400 | Sorafenib 400/400
Started | 3 | 5 | 0
Completed | 3 | 5 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase I
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 44 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities
Description: Number of dose limiting toxicities and number with adverse events.
  Dose-escalation schedule comprising 6 to 12 patients (see schema). This sample size is based on a traditional 3+3 cohort design with escalating doses of sorafenib in combination with 50 Gy of conformal radiotherapy delivered in 25 fractions (200 cGy per fraction). Based on preclinical data regarding the radiobiology of sorafenib,33, 36 sorafenib will be initiated at a dose of 200 mg twice daily, followed by 200 mg Q AM/400 mg Q PM for the 2nd cohort, followed by 400 mg bid for the 3rd cohort. Since 400 mg bid is the well established MTD for sorafenib monotherapy in patients with renal cell carcinoma and hepatocellular carcinoma, the dose will not be escalated above this level even if DLT is not observed. Dose level escalation will be determined based on DLTs observed from initiation of sorafenib/RT until time of surgery.
Time Frame: Approximately 12 weeks
Measure: Number; unit: DLTs
Arm/Group | Sorafenib 200/200 | Sorafenib 200/400
Number analyzed (Participants) | 3 | 5
DLTs | 0 | 2

ADVERSE EVENTS:
Groups:
- Sorafenib 200/200: Dose level 1. Sorafenib 200 mg PO BID
- Sorafenib 200/400: Dose level 2. Sorafenib 200 mg PO Q AM and 400 mg PO Q PM
Arm/Group | Sorafenib 200/200 | Sorafenib 200/400
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/5
Other Adverse Events (participants affected / at risk) | 2/3 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib 200/200 (N=3) | Sorafenib 200/400 (N=5)
rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib 200/200 (N=3) | Sorafenib 200/400 (N=5)
perirectal abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand-Foot syndrome (Nervous system disorders) | 1 (1) | 1 (1) — Palmar-plantar erythrodesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less